CLINICAL TRIAL: NCT05048069
Title: Post-Marketing Surveillance of Safety and Effectiveness of Mucosta®SR Tab. in Korean Patients With Acute or Chronic Gastritis in Accordance With Korean Regulation, 'Standard for Re-examination of New Drugs'
Brief Title: Post-Marketing Surveillance of Safety and Effectiveness of Mucosta®SR Tab.
Acronym: MCTSRPMS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Korea Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: 037-402-00047
Record Dates: First submitted 2021-08-24; First posted 2021-09-17 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Acute Gastritis; Chronic Gastritis
MeSH Terms: interventions — rebamipide

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Mucosta®SR Tablets 150mg(Rebamipide) — adult patients with gastric mucosal lesions (erosion, bleeding, redness, and edema) of acute gastritis or acute exacerbation of chronic gastritis prescribed with Mucosta®SR Tab. according to the medical considerations of the investigator.

SUMMARY:
This PMS is a non-interventional, prospective, single-arm, multi-center surveillance in accordance with Korean regulation, 'Standard for Re-Examination of New Drugs'. This PMS is to assess the safety and effectiveness after administrating Mucosta®SR Tab. Each subject would be observed for 2 weeks from baseline, if possible. As this PMS is an observational study in practical medical environment, the subject's follow-up is recommended but not obligatory and must be left up to the judgment of the investigator.

DETAILED DESCRIPTION:
According to the "Standards for Re-examination of New Drugs, etc." of South Korea, this PMS is conducted in order to collect safety and efficacy information for patients prescribed with Mucosta®SR Tab. under actual conditions of treatment during the re-examination period of Mucosta®SR Tab. 150mg (Rebamipide)

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients with gastric mucosal lesions (erosion, bleeding, redness, and edema) in acute gastritis or acute exacerbation of chronic gastritis.
2. Patients prescribed with Mucosta®SR Tab. according to the medical considerations of the investigator.
3. Patients who have given a written informed consent to participation of this PMS and use of personal information after execution of the contract with the surveillance study site.

Exclusion Criteria:

1. Patients with prior history of prescription with Mucosta®SR Tab.
2. Patients with hypersensitivity to Rebamipide or its component ingredients.
3. Patients deemed not suitable for surveillance enrollment according to investigator's medical judgment

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with gastric mucosal lesions (erosion, bleeding, redness, and edema) of acute gastritis or acute exacerbation of chronic gastritis prescribed with Mucosta®SR Tab. according to the medical considerations of the investigator.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2021-10-07 (Actual); Primary Completion 2024-12-15 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Overall clinical improvement | at 2 weeks of treatment
  Improved, No change, Worse The effective rate is defined as the percentage of subjects classified as 'Improved'.
the incidence rate and the number of cases for adverse events (AEs) | Safety information that occurred from the first administration to 3 days after discontinuation will be collected.

SECONDARY OUTCOMES:
Endoscopic improvement rate | at baseline and 2 weeks
  If upper GI endoscopy is performed at baseline and follow-up visits, the erosion score will be assessed and endoscopic improvement rate at 2 weeks will be evaluated. Endoscopic improvement rate is defined as ≥50% reduction of the erosion score.
Gastric symptoms | at baseline and 2 weeks
  Presence and type of gastric symptoms at baseline and 2 weeks will be collected.

CONTACTS AND LOCATIONS:
Locations (1):
- Soon Chun Hyang University Hospital Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No